CLINICAL TRIAL: NCT04814472
Title: A Two-Part, Open-Label, Crossover, Bioavailability Study Comparing Tablet and Oral Solution Formulations of BLD-0409 in Healthy Volunteers
Brief Title: Healthy Volunteer Study Comparing Tablet and Oral Solution Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blade Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B-0409-102
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Relative Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Solution vs. Tablet Formulation (Experimental): There will be 3 treatments, each single dose administered based on the treatment sequence with at least a 3 day washout between treatments:
  Treatment A: 750 mg BLD-0409 oral solution formulation (solution) under fasting conditions.
  Treatment B: 750 mg BLD-0409 tablet formulation (3 x 250 mg tablets) under fasting conditions.
  Treatment C: 750 mg BLD-0409 tablet formulation (3 x 250 mg tablets) under fed conditions.
  Interventions: Drug: BLD-0409
- Tablet Formulation Dose Proportionality (Experimental): There will be 4 treatments, each single dose administered under fed conditions (standard meal) based on the treatment sequence with at least a 3 day washout between treatments:
  Treatment A: 250 mg BLD-0409 tablet formulation (1 x 250 mg tablet).
  Treatment B: 500 mg BLD-0409 tablet formulation (2 x 250 mg tablet).
  Treatment C: 750 mg BLD-0409 tablet formulation (3 x 250 mg tablet).
  Treatment D: 1000 mg BLD-0409 tablet formulation (4 x 250 mg tablet).
  Interventions: Drug: BLD-0409

INTERVENTIONS:
Drug: BLD-0409 — Randomized to active product.

SUMMARY:
A Two-Part, Open-Label, Crossover, Bioavailability Study Comparing Tablet and Oral Solution Formulations of BLD-0409 in Healthy Volunteers

DETAILED DESCRIPTION:
The study will evaluate safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of two oral formulations of BLD-0409, tablet and solution, in healthy volunteers (HV).

The study consists of two parts:

Part 1: A randomized, open-label, 3-period, 6-sequence, complete crossover study with at least 3-day washout between treatment periods comparing oral solution formulation to tablet formulation.

Part 2: A randomized, open-label, 4-period, 4-sequence, complete crossover study with at least 3-day washout between treatment periods evaluating single ascending doses of tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Age and Gender

1. Male and female participants 18-55 years of age (inclusive) at the time of signing the PICF.

   Diagnosis and disease characteristics
2. Participants must be in good general health, in the opinion of the Investigator, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening, and/or before administration of the initial dose of study drug.
3. Participants must have clinical laboratory values within normal ranges or < 1.2 times upper limit of normal (ULN) as specified by the testing laboratory.
4. Body mass index (BMI) 18 to ≤ 32 kg/m2.

   Reproductive Considerations
5. Use of acceptable contraception.
6. Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1. Females not of childbearing potential must be surgically infertile or post-menopausal (defined as cessation of regular menstrual periods for at least 12 months), confirmed by follicle-stimulating hormone (FSH) level > 40 mIU/mL at Screening.

   Informed Consent
7. Participants must provide signed informed consent prior to study entry and have the ability and willingness to attend and comply with the necessary visits at the study site.

Exclusion Criteria:

Participants meeting ANY of the following exclusion criteria are NOT eligible to be randomized into the study:

Medical Conditions

1. Recent (less than 6 weeks) wound, or presence of an ongoing non-healing skin wound.
2. Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will complete the study per protocol.
3. Active malignancy and/or history of malignancy in the past 5 years, with the exception of completely excised non-melanoma skin cancer or low grade cervical intraepithelial neoplasia.
4. Serious local or systemic infection within 1 month of Screening requiring antibiotic treatment or history of recurrent infections.
5. Surgery within the past 3 months prior to the first study drug administration determined by the Investigator to be clinically relevant.

   Diagnostic Assessments
6. Positive for human immunodeficiency virus (HIV) antibody or antigen.
7. Positive hepatitis C virus (HCV) antibody or positive hepatitis B surface antigen (HBsAg).
8. Systolic blood pressure (BP) > 150 mmHg or < 90 mmHg or diastolic BP > 90 mmHg or < 50 mmHg at Screening with one repeat allowed per the Investigator's discretion at Screening and Day -1 (Period 1).
9. Heart rate < 40 beats per minute (bpm) or > 100 bpm at Screening.
10. Prolonged QT interval corrected by Fridericia's formula (QTcF) (> 450 ms for males and > 470 ms for females), cardiac arrhythmia, or any clinically significant abnormality in the resting ECG, as judged by the Investigator.
11. Females with heavy menstruating cycles and borderline-low iron studies.

    Prior Therapy
12. All prescription and over the counter medications (including herbal medications), except for non-estrogen contraceptives, are prohibited within 7 days prior to the first study drug administration and throughout the entire duration of the study.
13. Any estrogen-containing products, e.g., contraceptives, patch, cream, implants within 14 days prior to the first study drug administration.

    Prior/Concurrent Clinical Study Experience
14. Administration of investigational product in another study within 30 days prior to the first study drug administration, or five half-lives, whichever is longer.

    Other Exclusions
15. Significant weight loss or gain between Screening and first study drug administration.
16. Blood donation or significant blood loss within 60 days prior to the first study drug administration.
17. Plasma donation within 7 days prior to the first study drug administration.
18. Females who are pregnant or breastfeeding.
19. Diets that could alter metabolism (i.e., high protein, Slim Fast®, Nutrisystem®, etc.) within 7 days prior first study drug administration.
20. History or presence of alcohol or drug abuse (including recreational marijuana use) within the 1 year prior to the first study drug administration, and unwillingness to be totally abstinent during the dosing period.
21. Positive urine drug screen/alcohol breath test at Day -1 (admission).
22. Intake of alcohol or caffeine-containing products from 48 hours before first study drug administration through the EOS visit.
23. Active smokers and users of nicotine-containing products.
24. Failure to satisfy the Investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-05-16 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Area under the drug concentration-time curve from time zero to the last measurable concentration (AUC0-last) | Up to 16 days
  Measured by plasma concentration
Maximum observed drug concentration (Cmax) | Up to 16 days
  Measured by plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Argent, MD, Principal Investigator — Scientia
Locations (1):
- Scientia Clinical Research, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No